CLINICAL TRIAL: NCT05141799
Title: Effectiveness of High-intensity Laser Therapy in De Quervain Tenosynovitis; a Prospective, Randomized, Controlled Study
Brief Title: Effectiveness of High-intensity Laser Therapy in De Quervain Tenosynovitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Emine Dundar Ahi, MD, Assistant Professor, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2/2020.K-061
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: De Quervain Disease
Keywords: Hand grip strength; high-intensity laser therapy; De Quervain Disease
MeSH Terms: conditions — De Quervain Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-intensity laser therapy (HILT) (Active Comparator): we will apply the HILT device to the most painful area of the wrist in two phases. In both phase I and phase II, the laser will be applied using continuous circular movements.
  The first three sessions (phase I) will be used to provide analgesic effects at an intermittent phase, applying a 75 sec, 8 W, 6 J/cm2 treatment for a total of 150 J of energy. The subsequent six sessions (phase II) will provide a biostimulatory effect at a continuous phase, applying a 30 sec, 6 W, 120 to 150 J/cm2 treatment. The HILT will be applied for a total of nine treatment sessions over a period of three consecutive weeks.
  Interventions: Device: high intensity laser therapy
- sham HILT (Sham Comparator): We will apply the HILT device to the most painful area of the wrist by using continuous circular movements, but the laser instrument will switched off during applications. The sham HILT will be applied for a total of nine treatment sessions over a period of three consecutive weeks.
  Interventions: Device: high intensity laser therapy

INTERVENTIONS:
Device: high intensity laser therapy — Laser treatment is noninvasive and painless and can be easily administered in therapy units for a wide range of conditions. High-intensity laser therapy (HILT) has gained importance for the treatment of different kinds of sports injuries such as tendon injuries, contusions, and muscle spasms.

SUMMARY:
68 De Quervain tenosynovitis(MPS) diagnosed patients will be randomly divided into 2 groups. To groups; splinting+exercise+high-intensity laser therapy (HILT) and splinting+exercise+sham HILT will be applied. Visual anolog scale (VAS) scores, quick Disabilities of the Arm, Shoulder, and Hand (QDASH) questionnaire and Hand grip strength measurements of the patients before-after treatment will be recorded and will be evaluated statistically.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with unilateral De Quervain tenosynovitis 18-65 years old

Exclusion Criteria:

* pain history of less than four weeks,
* upper extremity entrapment neuropathy,
* major psychiatric disease,
* upper extremity surgical treatment history,
* malignancy history,
* chronic rheumatic disease,
* cervical radiculopathy,
* cervical myelopathy,
* local corticosteroid injection prior to De Quervain tenosynovitis and receiving physical therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
quick Disabilities of the Arm, Shoulder, and Hand (QDASH) questionnaire | 5 Minutes
  The QDASH is a self-reported questionnaire that measures the physical functions and symptoms of patients with upper limb problems. It includes 11 items from the DASH survey, and to calculate the QDASH score, atleast 10 of the 11 items should be answered. Each item contains five answer options, and the total score of the scale is calculated from the individual item scores (0=no disability and 100=the most serious disability). The first eight items of the QDASH questionnaire measure the patient's daily life function and social activity limitations. The ninth question assesses the pain intensity, and the 10th question evaluates the feeling of "pins and needles" in the upper extremity. The last question is designed to evaluate the sleep problem due to pain.
JAMAR hydraulic hand dynamometer | 2 minutes
  Hand grip strength measurements will take with a JAMAR hydraulic hand dynamometer (Lafayette Instrument, Lafayette, IN, USA) are known to provide reliable results and these measurements will be obtain while the patient will stand with a full extension of the elbow and wrist. Each patient will be asked to squeeze the dynamometer with full force for a maximum of three seconds. First on the healthy side and then on the effected side, three measurements will be taken, and the averages will be obtain.

SECONDARY OUTCOMES:
visual analog scale (VAS) | 10 Seconds
  Visual anolog scale (VAS) A Visual Analogue Scale (VAS) is a horizontal line, 100 mm in length measurement instrument that tries to measure the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Dundar Ahi, assist prof, Principal Investigator — Kocaeli University
Locations (1):
- Private Medar Hospital, Kocaeli, Golcuk, Turkey (Türkiye)